CLINICAL TRIAL: NCT04474314
Title: A Phase 2b Study to Evaluate the Safety and Efficacy of IMR-687 in Subjects With Sickle Cell Disease
Brief Title: A Study of IMR-687 in Subjects With Sickle Cell Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A recently conducted Interim analysis of IMR-SCD-301 demonstrated that while IMR-687 was generally well-tolerated, it failed to meet its primary efficacy endpoint. So, the sponsor has decided to discontinue this study.
Sponsor: Cardurion Pharmaceuticals, Inc. (Industry)
Collaborators: Imara, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IMR-SCD-301; 2019-004471-39 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-07-16 (Actual); Results first posted 2023-10-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Higher dose IMR-687 (Experimental): Oral administration of once daily IMR-687
  Interventions: Drug: IMR-687
- Lower Dose IMR-687 (Experimental): Oral administration of once daily IMR-687
  Interventions: Drug: IMR-687
- Placebo (Placebo Comparator): Oral administration of once daily Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IMR-687 — Oral administration of once daily IMR-687
  Arms: Higher dose IMR-687; Lower Dose IMR-687
Drug: Placebo — Oral administration of once daily Placebo
  Arms: Placebo

SUMMARY:
A Study to Evaluate the Safety and Efficacy of IMR-687 in Subjects with Sickle Cell Disease

DETAILED DESCRIPTION:
A phase 2b, randomized, double-blind, placebo-controlled, multicenter study of subjects with sickle cell disease (SCD; homozygous sickle hemoglobin [HbSS], sickle-β0 [HbSβ0] thalassemia, or sickle-β+ [HbSβ+] thalassemia) to evaluate the safety and efficacy of the phosphodiesterase type 9 (PDE9) inhibitor, IMR-687, administered once daily (qd) for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of SCD (HbSS, HbSB0 thalassemia, or HbSB+ thalassemia)
2. Hemoglobin of >5.5 and <10.5 g/dL; Hb values within 21 days post-transfusion will be excluded.
3. Subjects must have had at least 2 and no more than 12 documented episodes of VOCs in the past 12 months at the time of informed consent signing and at randomization (Day 1).
4. Subjects receiving HU must have received it continuously for at least 6 months prior to signing informed consent, and must have been on a stable dose for at least 3 months prior to signing the informed consent, with no anticipated need for dose adjustments during the study including the screening period, in the opinion of the investigator.
5. Female subjects must not be pregnant or breastfeeding and be highly unlikely to become pregnant. Male subjects must be unlikely to impregnate a partner.
6. Must be willing and able to complete all study assessments and procedures, and to communicate effectively with the investigator and site staff.

Exclusion Criteria:

1. Hospital discharge for sickle cell crisis or other vaso-occlusive event within the 4 days prior to randomization (Day 1).
2. Subjects participating in a chronic/prophylactic RBC transfusion program (i.e., regularly scheduled RBC transfusions); any transfusions within 21 days of screening or baseline Hb measurements
3. Subjects with HbF >25% at screening.
4. Significant kidney disease (eGFR <45mL/min) and liver dysfunction: alanine aminotransferase or aspartate aminotransferase >3x upper limit of normal.
5. Body mass index (BMI) <17.0 kg/m2 and a total body weight <45 kg; or a BMI >35 kg/m2.
6. Subjects with known active hepatitis A, hepatitis B, or hepatitis C, with active or acute event of malaria, or who are known to be positive for human immunodeficiency virus (HIV).
7. Stroke requiring medical intervention within 24 weeks prior to randomization (Day 1).
8. Prior exposure to IMR-687.
9. Subjects taking direct acting oral anti-coagulants (apixaban, dabigatran, rivaroxaban, edoxaban, or ticagrelor) or taking warfarin unless they stopped the treatment at least 28 days prior to randomization (Day 1).
10. A history of use of crizanlizumab (Adakveo®) or voxelotor (Oxbryta®) within 6 months prior to signing the informed consent.
11. Receipt of erythropoietin, luspatercept (Reblozyl®)or other hematopoietic growth factor treatment within 3 months of signing the ICF or anticipated need for such agents during the study.
12. Prior gene therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Attie, MD, Study Director — Imara, Inc.
Locations (49):
- United States (14):
  - University of Alabama at Birmingham School of Medicine - 1917 Clinic, Birmingham, Alabama
  - Arkansas Primary Care Clinic, Little Rock, Arkansas
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Center For Inherited Blood Disorders, Santa Ana, California
  - The Oncology Institute Long Beach, Whittier, California
  - University of Connecticut Health Main Building, Farmington, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - The University of Illinois at Chicago College of Medicine, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Weill Cornell Medicine - Center for Blood Disorders, New York, New York
  - Baylor Scott & White Medical Center-Temple, Temple, Texas
  - Virginia Commonwealth University Health - Ambulatory Care Center, Richmond, Virginia
- Ghana (2):
  - Korle Bu Teaching Hospital, Accra
  - Kintampo Health Research Centre, Kintampo
- Greece (3):
  - Laiko General Hospital of Athens, Athens, Attica
  - University General Hospital of Patras, Pátrai
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Italy (5):
  - Azienda Ospedaliero - Universitaria San Luigi Gonzaga, Turin, Orbassano
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma, Rome
  - Ente Ospedaliero Ospedali Galliera, Genoa
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello, Palermo
- Kenya (3):
  - Kenya Medical Research Institute - Kisumu, Kisumu, Nyanza
  - Gertrude's Children's Hospital, Nairobi
  - The Centre for Respiratory Diseases Research - Kenya Medical Research Institute, Nairobi
- Lebanon (3):
  - Hopital Nini, Tripoli, North Governorate
  - American University of Beirut Medical Center, Beirut
  - Chronic Care Center, Hazmiyeh
- Hôpital d'Enfants Rabat, Rabat, Morocco
- Hagaziekenhuis Van Den Haag - Leyweg, The Hague, South Holland, Netherlands
- Sultan Qaboos University Hospital, Muscat, Oman
- Centre National De Transfusion Sanguine - Du Senegal, Dakar, Senegal
- Tunisia (4):
  - Hedi Chaker Hospital, Sfax
  - Centre Hôpital Universitaire Farhat Hached, Sousse
  - Centre National de Greffe de la Moelle Osseuse, Tunis
  - Hospital Aziza Othmana, Tunis
- Uganda (5):
  - Jinja Regional Referral Hospital, Jinja
  - Uganda Cancer Institute, Kampala
  - Makerere University College of Health Sciences, Kampala
  - Joint Clinical Research Center - Lubowa, Kampala
  - Infectious Diseases Research Collaboration - Tororo, Tororo
- United Kingdom (6):
  - University Hospitals Bristol NHS Foundation Trust, Bristol, England
  - University College London Hospitals NHS, London, England
  - Guy's and Saint Thomas' NHS Foundation Trust, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Manchester University NHS Foundation Trust, Manchester, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Higher Dose IMR-687 | Lower Dose IMR-687 | Placebo
Started | 49 | 34 | 32
Completed | 2 | 6 | 8
Not Completed | 47 | 28 | 24

BASELINE CHARACTERISTICS:
Population: Intent to Treat Analysis set
Groups:
- Total: Total of all reporting groups
Arm/Group | Higher Dose IMR-687 | Lower Dose IMR-687 | Placebo | Total
Number analyzed (Participants) | 49 | 34 | 32 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.0 (7.91) | 27.9 (8.44) | 26.2 (9.27) | 26.2 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 14 | 14 | 64
  Male | 13 | 20 | 18 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 34 | 15 | 20 | 69
  White | 6 | 10 | 10 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 9 | 9 | 2 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 3 | 1 | 1 | 5
  Ghana | 11 | 2 | 8 | 21
  Kenya | 5 | 4 | 4 | 13
  Oman | 1 | 4 | 0 | 5
  Greece | 0 | 2 | 1 | 3
  Lebanon | 0 | 4 | 3 | 7
  Morocco | 5 | 2 | 3 | 10
  Senegal | 4 | 2 | 1 | 7
  Uganda | 16 | 8 | 5 | 29
  Tunisia | 1 | 3 | 4 | 8
  United States | 3 | 2 | 2 | 7
BMI [Mean (Standard Deviation); unit: kg/m^2] | 21.04 (3.571) | 21.03 (3.451) | 21.10 (2.794) | 21.06 (3.308)
HbF [Mean (Standard Deviation); unit: % of HbF] — Population: 1 participant in the high dose group was missing Baseline HbF
  % of HbF
    number analyzed (Participants) | 48 | 34 | 32 | 114
    (all) | 11.51 (7.775) | 10.16 (5.453) | 11.16 (4.903) | 11.01 (6.384)

OUTCOME MEASURES:

1. Primary Outcome: Effect on the Incidence of Vaso-occlusive Crises (VOCs)
Description: Annualized rate of VOCs. For each subject, the total number of VOCs on treatment were divided by the time on treatment divided by 52 weeks. The median was then summarized.
Time Frame: Baseline to Week 52
Population: ITT Analysis set
Measure: Median (Inter-Quartile Range); unit: VOCs/weeks/52
Arm/Group | Higher Dose IMR-687 | Lower Dose IMR-687 | Placebo
Number analyzed (Participants) | 47 | 33 | 32
VOCs/weeks/52 | 2.32 [1.02 to 5.51] | 1.20 [0.00 to 3.90] | 2.48 [0.51 to 5.03]

2. Primary Outcome: Proportion of Patients With Adverse Events and Serious Adverse Events
Description: Incidence of Adverse Events Incidence of Serious Adverse Events
Time Frame: Baseline to Week 56
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Higher Dose IMR-687 | Lower Dose IMR-687 | Placebo
Number analyzed (Participants) | 47 | 33 | 32
Participants
  Number of participants with Treatment-Emergent Adverse Events | 40 | 29 | 28
  Number of participants with Treatment Emergent Serious Adverse Events | 17 | 12 | 12

ADVERSE EVENTS:
Time Frame: 56 Weeks
Arm/Group | Higher Dose IMR-687 | Lower Dose IMR-687 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 17/47 | 12/33 | 12/32
Other Adverse Events (participants affected / at risk) | 38/47 | 29/33 | 24/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Dose IMR-687 (N=47) | Lower Dose IMR-687 (N=33) | Placebo (N=32)
Sickle Cell Anemia with Crisis (Blood and lymphatic system disorders) | 12 | 9 | 10
Anaemia (Blood and lymphatic system disorders) | 3 | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 2 | 1 | 2
Malaria (Infections and infestations) | 1 | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Higher Dose IMR-687 (N=47) | Lower Dose IMR-687 (N=33) | Placebo (N=32)
Headache (Nervous system disorders) | 12 | 9 | 7
Sickle Cell Anaemia with Crisis (Blood and lymphatic system disorders) | 12 | 9 | 10
Nausea (Gastrointestinal disorders) | 11 | 7 | 1
Dizziness (Nervous system disorders) | 10 | 3 | 2
Vomiting (Gastrointestinal disorders) | 9 | 6 | 0
Malaria (Infections and infestations) | 6 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04474314/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/14/NCT04474314/SAP_001.pdf